CLINICAL TRIAL: NCT07072884
Title: An Open-Label Study to Assess the Safety and Efficacy of GC012F in Patients With Autoimmune Diseases
Brief Title: GC012F in Patients With Autoimmune Diseases
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Qiong Fu (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Qiong Fu, Chief Physician of Rheumatology, RenJi Hospital
Organization: RenJi Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24105/D8318N00001
Record Dates: First submitted 2025-06-18; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-03

CONDITIONS: Systemic Sclerosis (SSc); Idiopathic Inflammatory Myopathy (IIM)
MeSH Terms: conditions — Scleroderma, Systemic; Myositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3.0×10^5 CAR-T cells/kg (Experimental)
  Interventions: Drug: GC012F injection

INTERVENTIONS:
Drug: GC012F injection — Subjects who meet the CAR-T cell infusion criteria will receive GC012F Injection infusion within 48-72 hours after completion of lymphodepleting preconditioning.

SUMMARY:
This is an open-label, early exploratory main clinical study to evaluate the safety and efficacy of GC012F Injection in subjects with autoimmune diseases (AID), as well as to assess its pharmacokinetic (PK) and pharmacodynamic (PD) profiles.

DETAILED DESCRIPTION:
This study consists of the following periods: screening period, apheresis day, baseline period, lymphodepleting preconditioning period, GC012F infusion, safety and efficacy follow-up period, and long-term follow-up period.

Eligible subjects will undergo apheresis and will receive the infusion following the manufacture of the chimeric antigen receptor T cell (CAR-T) product. Prior to CAR-T cell infusion, subjects will receive lymphodepleting preconditioning and will be assessed before infusion. Subjects who meet the criteria for cell infusion will receive CAR-T cell infusion, and the infusion dose for the same group or subsequent study groups may be adjusted based on safety and clinical efficacy. In this study, the CAR-T cell infusion dose is set as follows: one target dose group (Dose Group 1): 3.0×10^5 CAR-T cells/kg, and one alternative dose group (Dose Group -1): 2.0×10^5 CAR-T cells/kg or 1.0×10^5 CAR-T cells/kg, with a total of 15 evaluable subjects to be enrolled. Among them, 6 subjects will be enrolled during the dose-limiting toxicity (DLT) observation stage, and 9 subjects will be enrolled during the expansion stage. This study does not establish separate cohorts for different indications (systemic sclerosis [SSc] or idiopathic inflammatory myopathies [IIM]). Eligible subjects will receive a single infusion of GC012F Injection. After all 6 subjects in the DLT observation stage have completed DLT observation, all clinical study data collected during the DLT observation stage (primarily safety data) will be assessed. If no more than 1 out of the 6 subjects experiences a DLT, 9 additional subjects will be enrolled in the dose expansion stage. If 2 subjects experience a DLT, the investigators and partner will discuss and decide whether to explore a lower dose group (Dose Group -1).

After CAR-T cell infusion, subjects will be followed up for safety, cellular expansion and persistence, and efficacy until 672 days (96 weeks) after infusion, or until the subject withdraws from the study and declines further follow-up, death, withdrawal of informed consent, or loss to follow-up, whichever occurs first.

Leukapheresis: Only subjects who have completed screening and fully meet the eligibility criteria may be enrolled. Mononuclear cells will be collected from the enrolled subjects and transported to a Good Manufacturing Practice (GMP)-compliant manufacturing workshop for cell preparation.

Lymphodepleting preconditioning: After confirming that the cells have passed quality control and met the release criteria, the investigator will determine whether to initiate lymphodepleting preconditioning based on the subject's condition on Day -5 prior to GC012F Injection infusion. The preconditioning will last for a total of 3 days (Days -5, -4, and -3 or Days -4, -3, and -2). The recommended preconditioning regimen is as follows:

1. Fludarabine 30 mg/m^2/day, via intravenous infusion for 3 days;
2. Cyclophosphamide 300 mg/m^2/day, via intravenous infusion for 3 days. GC012F Injection infusion: Subjects who meet the CAR-T cell infusion criteria will receive GC012F Injection infusion within 48-72 hours after completion of lymphodepleting preconditioning.

Safety and efficacy follow-up: Subjects who receive GC012F Injection infusion should continue with all subsequent post-infusion assessments.

The inpatient observation period should start from the infusion (Day 0) and continue for 14 days; hospitalization from Day 15 to Day 28 should follow local diagnosis and treatment guidelines. The window for the Day 4, Day 7 (Week 1), Day 10, and Day 14 (Week 2) visits is ±1 day; for the Day 28 (Week 4) visit, the window is +3 days. Within 12 weeks after GC012F Injection infusion, follow-up visits will be conducted every 28 days (4 weeks) ±7 days (1 week). From Weeks 12 to 48, follow-up visits will be conducted every 84 days (12 weeks) ±7 days (1 week). After Week 48, follow-up visits will be conducted every 6 months (24 weeks) ±14 days (2 weeks), until 672 days (96 weeks) after infusion, withdrawal of informed consent, withdrawal from the study with refusal to undergo subsequent follow-up, death, or loss to follow-up, whichever occurs first. Subjects who do not withdraw from the study prematurely within 672 days (96 weeks) will proceed to the long-term follow-up period. The end of this study is defined as 672 days (96 weeks) after the last GC012F Injection infusion to the last subject.

Long-term follow-up: Subjects who do not withdraw from the study prematurely within 672 days (96 weeks) after infusion will proceed to the long-term follow-up period, which will continue until withdrawal of informed consent, withdrawal from the study with refusal to undergo subsequent follow-up, death, loss to follow-up, or 15 years after cell infusion, whichever occurs first. During this period, the primary focus will be on the collection of serious adverse events related to GC012F Injection. From Years 3 to 5 post-infusion, subjects will undergo follow-up every six months for replication competent lentivirus (RCL) and lentiviral integration site testing, and disease assessment-related examinations. From Years 6 to 15 post-infusion, subjects are required to undergo annual follow-up for RCL testing, lentiviral vector integration site testing, and disease assessment-related examinations.

Withdrawal visit: Subjects who withdraw from the study will undergo a withdrawal visit as specified. If a subject has initiated a new treatment prior to the withdrawal visit, details regarding the diagnostic basis for disease activity and the treatment process should be documented in chronological order unless the subject withdraws consent. There is no need to repeat the efficacy assessment at the withdrawal visit if it occurs within 4 weeks after the last two consecutive efficacy assessments. Other assessments do not need to be repeated if they are conducted within 2 weeks after the last assessment.

ELIGIBILITY:
Inclusion Criteria:

Only subjects who meet all of the following inclusion criteria prior to enrollment are eligible for this study. In addition, subjects should meet the relevant inclusion criteria for each indication as specified in the corresponding section of each sub-study protocol.

1. The subject or legal representative voluntarily signs the written informed consent form (ICF) personally, and is willing and able to comply with study procedures;
2. Aged 18 to 70 years (inclusive) at the time of signing the informed consent form, male or female;
3. Willing to adhere to study-specific contraception requirements until 2 years after infusion or until two consecutive flow cytometry tests indicate that CAR-T cells are no longer present in females of childbearing potential and male subjects (whichever occurs later);
4. Screening laboratory test results must meet the following criteria (except for indicators related to the diseases under study):

   1. Neutrophil count ≥ 1.0 × 10^9/L; hemoglobin ≥ 80 g/L; platelet count ≥ 50 × 10^9/L;
   2. Alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN); aspartate aminotransferase (AST) ≤ 3 × ULN (unless ALT and/or AST increase is assessed by the investigator as related to IIM); total bilirubin < 2 × ULN (for subjects with Gilbert's syndrome, direct bilirubin ≤ 1.5 × ULN);
   3. Creatinine clearance ≥ 60 mL/min, or estimated glomerular filtration rate (eGFR) ≥ 45 mL/min/1.73 m^2;
   4. Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, and prothrombin time (PT) ≤ 1.5 × ULN;
   5. Left ventricular ejection fraction (LVEF) ≥ 50% as determined by echocardiogram, with no evidence of pericardial effusion.
5. Women of childbearing potential must:

   1. Have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result at screening as confirmed by the investigator;
   2. Agree to avoid breastfeeding during the study period and until at least 2 years after infusion of GC012F Injection, or until two consecutive flow cytometry tests indicate that CAR-T cells are no longer present (whichever occurs later).
6. Male subjects with sexual partners and female subjects of childbearing potential must agree to use highly effective contraception methods (e.g., oral contraceptives, intrauterine devices, or condoms) starting from screening and continuing for at least 2 years after GC012F Injection infusion or until two consecutive flow cytometry tests indicate that CAR-T cells are no longer present (whichever occurs later). Male subjects must agree to use condoms during any sexual contact with pregnant women or women of childbearing potential for at least 2 years after GC012F Injection infusion, even if they have undergone successful vasoligation.
7. The required venous access for collection can be set up, with no contraindications for leukapheresis.

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible for the study. In addition, subjects who meet the relevant exclusion criteria for each indication as specified in the corresponding section of each sub-study protocol must not be enrolled.

1. History of severe hypersensitivity or allergy;
2. Contraindications or hypersensitivity to fludarabine, cyclophosphamide, or any component of the investigational product;
3. Presence of the following cardiac disorders:

   1. New York Heart Association (NYHA) Class III or IV congestive heart failure;
   2. Myocardial infarction or coronary artery bypass grafting within 6 months prior to screening;
   3. History of clinically significant ventricular arrhythmia or unexplained syncope not caused by vasovagal reactions or dehydration, or corrected QT interval > 480 ms at screening;
   4. History of severe non-ischemic cardiomyopathy.
4. Any active malignancy or history of malignancy within 5 years prior to screening. The following are exceptions: early-stage tumors that have received curative treatment (carcinoma in situ or stage I tumors, non-ulcerative primary melanoma with a depth < 1 mm and no lymph node involvement), basal cell carcinoma of the skin, squamous cell carcinoma of the skin, thyroid carcinoma in situ or early-stage thyroid cancer that has received curative treatment, cervical carcinoma in situ, or breast cancer in situ that has received potentially curative treatment;
5. Clinically significant hemorrhage symptoms or a definite tendency to hemorrhage within 6 months prior to screening, such as hemorrhage of digestive tract and hemorrhagic gastric ulcer; hereditary or acquired hemorrhage or thrombotic tendencies (e.g., hemophilia, coagulation disorders, and hypersplenism); arterial or venous thrombotic events within 6 months prior to screening, such as cerebrovascular diseases (including cerebral hemorrhage and cerebral infarction), deep vein thrombosis and/or pulmonary embolism;
6. Any of the following test results is positive:

   1. Human immunodeficiency virus (HIV) antibody positive;
   2. Hepatitis B surface antigen (HBsAg) positive; or hepatitis B core antibody (HBcAb) positive with hepatitis B virus deoxyribonucleic acid (DNA) above the lower limit of detection of the assay;
   3. Hepatitis C virus (HCV) antibody positive with HCV ribonucleic acid (RNA) above the lower limit of detection of the assay;
   4. Syphilis antibody positive (confirmation by a confirmatory test for syphilis is required if necessary, such as fluorescent treponemal antibody-absorption test and Treponema pallidum particle agglutination assay).
7. Active tuberculosis or latent tuberculosis that has not received appropriate treatment prior to screening;
8. Severe underlying medical conditions, such as:

   1. Evidence of viral, bacterial, fungal, or other infections that are uncontrolled or need systemic intravenous treatment;
   2. Clear clinical evidence of dementia or altered mental status;
   3. Any other central nervous system disease or history of neurodegenerative diseases, such as epilepsy, seizure, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, and psychosis.
9. Prior therapy targeting cluster of differentiation (CD)19 and/or B-cell maturation antigen, or CAR-T product therapy targeting any antigen;
10. Thymectomy within 12 months prior to signing the ICF;
11. Treatment with CD20-targeted agents within 6 months prior to signing the ICF;
12. Receipt of other investigational products within 4 weeks prior to signing the ICF, or if the time from the last dose of a previous investigational product to the ICF signing date is still within 5 half-lives of that drug (whichever is longer);
13. Receipt of other monoclonal antibody drugs (e.g., infliximab, certolizumab pegol, golimumab, etanercept, abatacept, adalimumab, or tocilizumab) within 4 weeks prior to apheresis;
14. Receipt of cyclophosphamide within 4 weeks prior to apheresis;
15. Major surgery within 8 weeks prior to signing the ICF, or planned surgery during the study;
16. History of organ transplantation;
17. Pregnant women, breastfeeding women who do not agree to discontinue breastfeeding, or males and females who plan to conceive during the study or within 2 years after receiving study treatment;
18. Any condition, as determined by the investigator, that would interfere with the subject's full participation in the study, confound the study results, or render participation in the study not in the best interest of the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with dose-limiting toxicity (DLT) within 28 days after infusion. | 28 days after infusion.
Post-infusion adverse events and their proportion. | From the signing of informed consent through 672 days (96 weeks) after cell infusion or initiation of a new therapy, whichever occurs first.

SECONDARY OUTCOMES:
Chimeric antigen receptor T cell (CAR-T) levels in peripheral blood at each time point. | From the signing of informed consent through 672 days (96 weeks) after cell infusion or initiation of a new therapy, whichever occurs first.
Chimeric antigen receptor transgene levels in peripheral blood at each time point. | From the signing of informed consent through 672 days (96 weeks) after cell infusion or initiation of a new therapy, whichever occurs first.
Quantification of cytokines in peripheral blood at each time point. | From the signing of informed consent through 672 days (96 weeks) after cell infusion or initiation of a new therapy, whichever occurs first.
Quantification of immunoglobulins in peripheral blood at each time point. | From the signing of informed consent through 672 days (96 weeks) after cell infusion or initiation of a new therapy, whichever occurs first.
Changes in patient reported outcomes (PROs) from baseline at each time point: health assessment questionnaire disability index (HAQ-DI) . | From the signing of informed consent through 672 days (96 weeks) after cell infusion or initiation of a new therapy, whichever occurs first.
Changes in patient reported outcomes (PROs) from baseline at each time point: patient global activity assessment (PtGA). | From the signing of informed consent through 672 days (96 weeks) after cell infusion or initiation of a new therapy, whichever occurs first.

OTHER OUTCOMES:
Detection rate of CAR-T cell antibody after GC012F infusion. | From the signing of informed consent through 672 days (96 weeks) after cell infusion or initiation of a new therapy, whichever occurs first.
Changes in antibody concentrations resulting from previous vaccination. | From the signing of informed consent through 672 days (96 weeks) after cell infusion or initiation of a new therapy, whichever occurs first.
Detection rate of RCL after GC012F infusion. | From the signing of informed consent through 672 days (96 weeks) after cell infusion or initiation of a new therapy, whichever occurs first.

IPD SHARING:
Plan to Share IPD: No